CLINICAL TRIAL: NCT02876562
Title: Comparitive Evaluation of Modified Coronally Advanced Tunnel Collagen Matrix Versus Connective Tissue Graft for Root Coverage in Multiple Gingival Recessions-A Randomised Controlled Clinical Trial
Brief Title: A Comparision of Collagen Matrix and Connective Tissue Graft With Modified Coronally Advanced Tunnel for Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_63804
Record Dates: First submitted 2016-07-28; First posted 2016-08-24 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2016-04

CONDITIONS: Gingival Recession
Keywords: Gingival Recession Coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- root coverage with collagen matrix (Experimental): evaluation of root coverage achieved by collagen matrix in conjunction with modified coronally advanced tunnel in patients with multiple gingival recession
  Interventions: Procedure: root coverage with collagen matrix
- root coverage with connective tissue graft (Active Comparator): evaluation of root coverage achieved by connective tissue graft in conjunction with modified coronally advanced tunnel in patients with multiple gingival recession
  Interventions: Procedure: root coverage with collagen matrix

INTERVENTIONS:
Procedure: root coverage with collagen matrix — the material used is a porcine derived native collagen matrix which serves an alternative to connective tissue graft. the material is 1.5 mm in thickness with a specific tissue surface to allow for cell migration and a fibrous outer layer. it has a resorption time of 6 months.

SUMMARY:
Recently porcine derived bioresorbable collagen matrices have shown predictable outcomes for augmenting keratinzed gingiva , improved wound healing, recession coverage in localized gingival recessions and multiple recession coverage.

However there are very few randomized controlled clinical trials in the literature that compare collagen matrix versus connective tissue graft in the management of multiple recession type defects. To the best of our knowledge there is only one randomized controlled trial that compares modified coronally advanced tunnel+connective tissue graft with collagen matrix in the management of multiple gingival recessions.

Thus aim of this study will be to compare the effectiveness of collagen versus CTG in the management of Millers class I and II multiple gingival recessions. The use of collagen matrix in combination with Modified Coronally Advanced Tunnel as a surgical technique will be compared for recession coverage.

DETAILED DESCRIPTION:
Gingival recession is defined as the displacement of the soft tissue margin apical to cementoenamel junction and it may affect single or multiple root surfaces. Gingival recessions are known to compromise esthetic appearance, hinder plaque control, and result in higher susceptibility to hypersensitivity and root caries.

It can be the result of different predisposing anatomic features such as thin gingival biotype, buccal prominence of teeth, lack of keratinized tissue, high frenal attachment, or patient related factors such as vigorous brushing or chronic gingival inflammation. Recessions may be localized or generalized. Alternatively they have been classified into four classes on the basis of extent. Miller's Class I and Class II recession defects mainly occur in multiple buccal areas and the main etiologic factors include trauma from tooth brushing. Miller's Class III and Class IV recessions usually involve the whole mouth and is often related to plaque associated chronic inflammatory periodontal disease. Because of their traumatic etiology, multiple recessions are more frequent.

It has been extensively demonstrated that in Miller's Class I and II single recessions, complete root coverage can be predictably achieved with various techniques. On the other hand, treatment of multiple adjacent gingival recessions is still a challenge for the clinician as in these cases the management of soft tissues becomes more difficult and the wound healing may be compromised by various factors such as width of avascular surface, limited blood supply, differences in the recession depth and position of the teeth. The ultimate goal of root coverage procedures is the complete coverage of the recession defect, with good esthetics and harmonious integration of the covering tissues and with minimal probing depths after treatment.

A variety of surgical procedures have been used to cover exposed root surfaces such as Laterally Positioned Flap, Coronally Advanced Flap, Modified Coronally Advanced Flap, Coronally Advanced Tunnel, Modified Coronally Advanced Tunnel, Subepithelial Connective Tissue Graft(SCTG), Acellular Dermal Matrix(ADMA) and Guided Tissue Regeneration.

Coronally advanced flap (CAF) and SCTG are the most predictable techniques, achieving up to 100% root coverage. CAF alone and with various modifications have been used widely and successfully. Studies have stated that SCTG has not only the highest percentage of mean root coverage but also least variability. In spite of its promising results, SCTG has its own limitations, such as lack of graft availability, need for a second surgical site, proximity to palatine neurovascular complex and unesthetic contour at the recipient site. In some cases, harvesting connective tissue may be difficult in the presence of a flat palatal profile or if thickness of masticatory mucosa appears too thin. The additional chair time must also be considered and compared with that needed to perform a CAF alone. But it has been noted in various studies that CAF alone is not as effective as CAF with CTG, which leads to the attempt of finding an alternative to CTG with all the benefits and none of its drawbacks.

Variants such as membranes, biologic modifiers, and allografts have been developed and tested as substitutes for CTG. Collagen matrix(CM), composed of non-crosslinked porcine collagen, is one such substitute. The matrix is intended to support 3D soft tissue regeneration by favouring blood clot stabilization and early vascularization by its excellent tissue integration. It consists of a superficial cell occlusive layer, and a deeper porous layer. The primary importance of CM lies in that it functions almost as well as CTG in procedures for root coverage and those performed to increase the dimensions of keratinized gingiva, at the same time avoiding all the negatives of the latter. The additional advantages of CM is its influence on the healing cascade and reduced scar retraction. Also it leads to increased thickness of keratinized gingiva thus remedying one of the etiolgical factors of gingival recession. The advent of such materials could have a revolutionary impact within the field of periodontics.

But this merits further research and study in this direction to clarify the position of collagen matrices as a substitute for CTG in periodontal plastic surgeries. Therefore the need for this study is to evaluate the efficacy of collagen matrix as a definitive alternative for CTG and if it will be able to supplant CTG as the most effective method to treat gingival recessions.

Tunnel technique in perioplastic surgery was first introduced by Allen in 1994 , and followed by modifications by Zabalegui(1999), Modified Coronally Advanced Tunnel(MCAT), and Microsurgical CAT. All these techniques have shown remarkable success with root coverage. MCAT technique has certain advantages over CAF/ Modified CAF as the vascular supply of the coronally advanced component is not compromised due to avoidance of vertical/ horizontal incisions.

Recently porcine derived bioresorbable collagen matrices have shown predictable outcomes for augmenting keratinzed gingiva, improved wound healing, recession coverage in localized gingival recession and multiple recession coverage.

However there are very few randomized controlled clinical trials in the literature that compare collagen matrix versus CTG in the management of MRTDs. To the best of our knowledge there is only one RCT that compares MCAT+CTG with MCAT+CM in the management of multiple gingival recessions.

Thus aim of this study will be to compare the effectiveness of collagen versus CTG in the management of Millers class I and II multiple gingival recessions. The use of collagen matrix in combination with Modified Coronally Advanced Tunnel as a surgical technique will be compared for recession coverage.

ELIGIBILITY:
Inclusion Criteria:• Multiple Millers class I and II or combined class I and II recession defects in maxillary or mandibular arches

* Age >/= 18
* Patients with thick gingival biotypes(>0.8mm)24
* Patients with healthy or treated periodontal conditions.8
* Patients willing to participate in the study.8
* Absence of uncontrolled medical conditions25
* Full mouth plaque score </= 10%(O'Leary 1972)
* Patients with esthetic concerns.

Exclusion Criteria:

* • Pregnant or lactating females 8

  * Tobacco smoking26
  * Uncontrolled medical conditions25
  * Untreated periodontal conditions
  * Use of systemic antibiotics in the past 3 months
  * Patients treated with any medication known to cause gingival hyperplasia8
  * Drug and alcohol abuse8
  * Recession defects associated with occlusal interferences, pulpal pathology, caries/demineralization, restorations and deep abrasions( step>2mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
gingival recession depth | 6 months
gingival recession width | 6 months
complete root coverage | 6 months
clinical attachment level | 6 months
keratinized tissue width | 6 months
probing depth | 6 months

SECONDARY OUTCOMES:
plaque index | 6 months
gingival bleeding index | 6 months
gingival index | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya College of Dental Sciences, Bangalore, Karnataka, India